CLINICAL TRIAL: NCT01979445
Title: A Study of the Transition From Cangrelor to Clopidogrel or Prasugrel in Patients With Coronary Artery Disease.
Brief Title: Cangrelor to Clopidogrel or Prasugrel Transition Study
Acronym: BRIDGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MDCO-CAN-13-02
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease | interventions — cangrelor; Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Prasugrel 30 Min After Cangrelor (Experimental): Prasugrel 60 milligram (mg) administered orally 30 min after the discontinuation of cangrelor infusion on Day 1 (2.5 hours [hrs] after initiation of cangrelor infusion).
  Interventions: Drug: Cangrelor; Drug: Prasugrel
- Clopidogrel Within 5 Min After Cangrelor (Experimental): Clopidogrel 600 mg administered orally within 5 min after the discontinuation of the cangrelor infusion on Day 1 (2 hrs after initiation of cangrelor infusion).
  Interventions: Drug: Cangrelor; Drug: Clopidogrel
- Clopidogrel 1.5 Hrs During Cangrelor (Experimental): Clopidogrel 600 mg administered orally 1.5 hrs after the initiation of cangrelor infusion on Day 1.
  Interventions: Drug: Cangrelor; Drug: Clopidogrel
- Clopidogrel 1 Hr During Cangrelor (Experimental): Clopidogrel 600 mg administered orally 1 hr after the initiation of cangrelor infusion on Day 1.
  Interventions: Drug: Cangrelor; Drug: Clopidogrel

INTERVENTIONS:
Drug: Cangrelor — Cangrelor intravenously (IV) administered as a 30 microgram (µg)/kilogram (kg) bolus, followed by 4 µg/kg/min infusion for 2 hrs on Day 1.
Drug: Clopidogrel — Clopidogrel 600 mg single oral dose
  Arms: Clopidogrel 1 Hr During Cangrelor; Clopidogrel 1.5 Hrs During Cangrelor; Clopidogrel Within 5 Min After Cangrelor
Drug: Prasugrel — Prasugrel 60 mg single oral dose
  Arms: Prasugrel 30 Min After Cangrelor

SUMMARY:
There are two separate objectives in this study:

1. To demonstrate the pharmacodynamic (PD) profile when participants treated with cangrelor are switched to oral prasugrel 60 mg administered 30 minutes (min) after cangrelor infusion is discontinued
2. To demonstrate the PD profile when participants treated with cangrelor are switched to oral clopidogrel 600 mg administered during or immediately after cangrelor infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 and less than 75 years of age, of either sex, and of any race.
2. Stable CAD defined by the following criteria:

   1. Previous myocardial infarction defined by admission to the hospital with elevation of markers of injury or the presence of pathologic Q-waves on at least 2 contiguous electrocardiogram (ECG) leads.

      or
   2. Previous revascularization by percutaneous coronary intervention or coronary artery bypass graft, and
   3. Treatment with aspirin 81 mg daily.

Exclusion Criteria:

1. Known intolerance or contraindication to cangrelor or prasugrel, or any ingredients of the respective formulation.
2. Any antiplatelet (other than aspirin) or anticoagulant medication within the previous 30 days.
3. Acute coronary syndrome within the previous 12 months.
4. History of bleeding diathesis or known coagulopathy such as; impaired hemostasis; known international normalized ratio (INR) >1.5; past or present bleeding disorder (including congenital bleeding disorders, such as, von Willebrand's disease or hemophilia), acquired bleeding disorders, and unexplained clinically significant bleeding disorders; thrombocytopenia (platelet count less than 100,000/microliter [µL]), or history of thrombocytopenia or neutropenia associated with clopidogrel.
5. Anemia (for example, hematocrit less than 35%).
6. Prior stroke (any type), prior cerebral arteriovenous malformation or intracranial aneurysm; recent (<1 month) trauma or major surgery (including bypass surgery).
7. Known or suspected pregnancy, or lactating females.
8. Known severe renal insufficiency (glomerular filtration rate less than 30 milliliter [mL]/min).
9. Inability to provide informed consent.
10. Moderate or severe hepatic impairment as per Investigator's discretion (elevation of liver function tests).
11. Inability to swallow oral medication at time of randomization.
12. Any clinically significant disease or condition affecting a major organ system, including but not limited to gastrointestinal, renal, hepatic, endocrinologic, broncho-pulmonary, neurological, or metabolic disease.
13. Any surgical or medical condition which, in the judgment of the Investigator, might interfere with the pharmacokinetics, distribution, metabolism, or excretion of the study drug (if applicable).
14. Treatment with other investigational medicinal products or devices within 30 days or 5 half-lives, whichever is longer, prior to the administration of the drug, or planned use of investigational medicinal products or devices.
15. Participants who, for any reason, are deemed by the Investigator to be inappropriate for this study, including participants who are unable to communicate or to cooperate with the Investigator.
16. Participant is the Investigator or his/her deputy, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.
17. Active pathological bleeding, or a history of transient ischemic attack.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2014-01-20 (Actual); Study Completion 2014-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Schneider, MD, Principal Investigator — University of Vermont Medical Center
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States

REFERENCES:
- [Result] Schneider DJ, Agarwal Z, Seecheran N, Gogo P. Pharmacodynamic Effects When Clopidogrel is Given Before Cangrelor Discontinuation. J Interv Cardiol. 2015 Oct;28(5):415-9. doi: 10.1111/joic.12229. Epub 2015 Sep 18. PMID 26381736

RESULTS

PARTICIPANT FLOW:
Groups:
- Prasugrel 30 Min After Cangrelor: Cangrelor intravenously (IV) was administered on Day 1 as a 30 microgram (μg)/kilogram (kg) bolus, followed by 4 μg/kg/minute (min) infusion for 2 hours (hrs).
  Prasugrel 60 milligram (mg) was administered on Day 1 as a single oral dose 30 min after the discontinuation of cangrelor infusion (2.5 hrs after initiation of cangrelor infusion).
- Clopidogrel Within 5 Min After Cangrelor: Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
  Clopidogrel 600 mg was administered on Day 1 as a single oral dose within 5 min after the discontinuation of the cangrelor infusion (2 hrs after initiation of cangrelor infusion).
- Clopidogrel 1.5 Hrs During Cangrelor: Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
  Clopidogrel 600 mg was administered on Day 1 as a single oral dose 1.5 hrs following the initiation of cangrelor infusion.
- Clopidogrel 1 Hr During Cangrelor: Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
  Clopidogrel 600 mg was administered on Day 1 as a single oral dose 1 hr following the initiation of cangrelor infusion.
Period: Overall Study
Arm/Group | Prasugrel 30 Min After Cangrelor | Clopidogrel Within 5 Min After Cangrelor | Clopidogrel 1.5 Hrs During Cangrelor | Clopidogrel 1 Hr During Cangrelor
Started | 3 | 3 | 6 | 3
Received at Least 1 Dose of Study Drug (Safety Population included all participants who received at least 1 dose of study drug.) | 3 | 3 | 6 | 3
ITT Population (Intent to treat (ITT) Population included all enrolled participants in the study.) | 3 | 3 | 6 | 3
Completed | 3 | 3 | 6 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received prasugrel or clopidgrel.
Groups:
- Prasugrel: Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
  Prasugrel 60 mg was administered on Day 1 as a single oral dose 30 min on Day 1 after the discontinuation of cangrelor infusion.
- Clopidogrel: Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs on Day 1.
  Clopidogrel 600 mg was administered on Day 1 as a single oral dose 1 and 1.5 hrs after the initiation of cangrelor infusion and within 5 min after the discontinuation of the cangrelor infusion.
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Clopidogrel | Total
Number analyzed (Participants) | 3 | 12 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (6.66) | 65.3 (6.18) | 64.7 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 12 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 12 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 12 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 12 | 15

OUTCOME MEASURES:

1. Primary Outcome: Extent of Preservation Of Platelet Inhibitory Effect After Transition From Cangrelor To Prasugrel Or Clopidogrel Compared With Effect Observed With Prasugrel Or Clopidogrel Alone
Description: A reference point for prasugrel or clopidogrel was chosen for comparison and designated at 6 or 5.5 hrs after the administration of prasugrel or clopidogrel as the reference for the effect of the oral drug. Platelet function was assessed using light transmittance aggregometry (LTA). LTA measures the aggregation or cross linking of platelets by fibrinogen and requires the activation of platelets plus the binding of fibrinogen. The extent of aggregation was expressed as % aggregation in response to 20 micromolar (μM) adenosine diphosphate (ADP) at 300 seconds (sec) (final/terminal aggregation response).
Time Frame: Day 1 at 5.5 or 6 hrs after administration of prasugrel or clopidogrel (reference) and Day 1 at 2.25, 2.5, 2.75, 3, 4, and 5.5 hrs after initiation of cangrelor infusion
Population: Participants treated with cangrelor and prasugrel or clopidogrel were used for the analysis and presentation of data.
Measure: Mean (Standard Deviation); unit: % aggregation
Groups:
- Prasugrel 30 Min After Cangrelor: Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
  Prasugrel 60 mg was administered on Day 1 as a single oral dose 30 min after the discontinuation of cangrelor infusion (2.5 hrs after initiation of cangrelor infusion).
Arm/Group | Prasugrel 30 Min After Cangrelor | Clopidogrel Within 5 Min After Cangrelor | Clopidogrel 1.5 Hrs During Cangrelor | Clopidogrel 1 Hr During Cangrelor
Number analyzed (Participants) | 3 | 3 | 6 | 3
% aggregation
  Prasugrel/Clopidogrel Reference (6 or 5.5 hrs) | 1.3 (1.5) | 21.7 (16.4) | 50.0 (16.8) | 50.3 (15.9)
  2.25 hrs | 16.3 (10.1) | 26.0 (7.9) | 22.2 (16.0) | 33.3 (7.5)
  2.5 hrs | 60.0 (7.5) | 49.7 (7.1) | 54.3 (11.7) | 62.0 (3.6)
  2.75 hrs | 63.3 (1.5) | 58.3 (7.4) | 56.8 (11.3) | 67.7 (1.2)
  3 hrs | 65.0 (2.0) | 56.0 (8.9) | 56.2 (16.4) | 65.0 (9.5)
  4 hrs | 16.3 (27.4) | 38.0 (31.7) | 51.2 (27.4) | 62.7 (8.5)
  5.5 hrs | 1.3 (1.5) | 26.7 (20.5) | NA (NA) — Per protocol, analysis was not performed at 5.5 hrs for this arm. | NA (NA) — Per protocol, analysis was not performed at 5.5 hrs for this arm.

2. Primary Outcome: Extent Of Preservation Of Platelet Inhibitory Effect Of Cangrelor Treatment After Prasugrel Or Clopidogrel Compared To Treatment With Cangrelor Alone
Description: A reference point for cangrelor was chosen for comparison and designated as the administration time of prasugrel 60 mg or clopidogrel 600 mg (2.5, 2, 1.5, or 1 hrs). Platelet function was assessed using LTA. LTA measures the aggregation or cross linking of platelets by fibrinogen and requires the activation of platelets plus the binding of fibrinogen. The extent of aggregation was examined using LTA and expressed as % aggregation in response to 20 μM ADP at 300 sec (final/terminal aggregation response).
Time Frame: Day 1 at 1, 1.5, 2, or 2.5 hrs after administration of prasugrel or clopidogrel (reference) and Day 1 at 1.75 and 2 hrs after initiation of cangrelor infusion
Population: Participants treated with cangrelor and prasugrel or clopidogrel were used for the analysis and presentation of data.
Measure: Mean (Standard Deviation); unit: % aggregation
Groups:
- Clopidogrel 1 Hr During Cangrelor: Clopidogrel 600 mg was administered on Day 1 as a single oral dose 1 hr following the initiation of cangrelor infusion.
  Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
Arm/Group | Prasugrel 30 Min After Cangrelor | Clopidogrel Within 5 Min After Cangrelor | Clopidogrel 1.5 Hrs During Cangrelor | Clopidogrel 1 Hr During Cangrelor
Number analyzed (Participants) | 3 | 3 | 6 | 3
% aggregation
  Cangrelor Reference (2.5, 2, 1.5, or 1 hrs) | 60.0 (7.5) | 0 (0) | 2.0 (3.5) | 3.0 (2.0)
  1.75 hrs | 0.3 (0.6) | 1.0 (1.0) | 1.8 (2.5) | 1.3 (0.6)
  2 hrs | 0.3 (0.6) | NA (NA) — Per protocol, analysis was not performed at 2 hrs for this arm. | 1.5 (2.0) | 2.3 (1.2)

3. Secondary Outcome: Extent of Preservation Of Platelet Inhibitory Effect After Transition From Cangrelor to Prasugrel Or Clopidogrel Compared With Effect Observed With Prasugrel Or Clopidogrel Alone Determined By VerifyNow P2Y12 Assay
Description: A reference point for prasugrel or clopidogrel was chosen for comparison and designated at 6 or 5.5 hrs after the administration of prasugrel or clopidogrel as the reference for the effect of the oral drug. Platelet function was assessed using the VerifyNow P2Y12 assay. The VerifyNow P2Y12 assay measures the aggregation or cross linking of platelets by fibrinogen and requires the activation of platelets plus the binding of fibrinogen. The extent of aggregation was assessed by platelet reaction units (PRU), determined by the VerifyNow P2Y12 assay. The VerifyNow P2Y12 assay is designed to directly measure the effects of drugs on the P2Y12 receptor, using prostaglandin E1 in addition to ADP to increase intraplatelet cyclic adenosine monophosphate (cAMP). Platelet reactivity was expressed in PRU.
Time Frame: as for outcome 1
Population: Participants treated with cangrelor and prasugrel or clopidogrel were used for the analysis and presentation of data.
Measure: Mean (Standard Deviation); unit: PRU
Groups:
- Clopidogrel Within 5 Min Post Cangrelor: Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
  Clopidogrel 600 mg was administered on Day 1 as a single oral dose within 5 min after the discontinuation of the cangrelor infusion (2 hrs after initiation of cangrelor infusion).
- Clopidogrel 1.5 Hrs During Cangrelor: Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
  Clopidogrel 600 mg administered on Day 1 as a single oral dose 1.5 hrs following the initiation of cangrelor infusion.
Arm/Group | Prasugrel 30 Min After Cangrelor | Clopidogrel Within 5 Min Post Cangrelor | Clopidogrel 1.5 Hrs During Cangrelor | Clopidogrel 1 Hr During Cangrelor
Number analyzed (Participants) | 3 | 3 | 6 | 3
PRU
  Prasugrel/Clopidogrel Reference (6 or 5.5 hrs) | 8.0 (8.7) | 159.0 (72.7) | 211.3 (66.8) | 197.3 (15.0)
  2.25 hrs | 76.7 (23.7) | 99.0 (27.6) | 90.3 (32.3) | 98.7 (19.6)
  2.5 hrs | 208.0 (30.2) | 220.7 (11.6) | 229.8 (24.6) | 206.3 (26.9)
  2.75 hrs | 225.7 (42.5) | 233.0 (21.7) | 255.8 (43.7) | 214.3 (11.9)
  3 hrs | 226.0 (28.5) | 215.7 (35.0) | 234.5 (34.2) | 212.7 (10.3)
  4 hrs | 77.0 (126.5) | 182.0 (82.3) | 215.5 (67.4) | 203.7 (11.2)
  5.5 hrs | 24.5 (34.6) | 155.0 (69.8) | NA (NA) — Per protocol, analysis was not performed for this arm at 5.5 hrs. | NA (NA) — Per protocol, analysis was not performed for this arm at 5.5 hrs.

4. Secondary Outcome: Extent of Preservation of Platelet Inhibitory Effect of Cangrelor Treatment After Prasugrel or Clopidogrel Compared to Treatment With Cangrelor Alone Determined By VerifyNow P2Y12 Assay
Description: A reference point for cangrelor was chosen for comparison and designated as the administration time of prasugrel 60 mg or clopidogrel 600 mg (2.5, 2, 1.5, or 1 hrs). Platelet function was assessed using the VerifyNow P2Y12 assay. The VerifyNow P2Y12 assay measures the aggregation or cross linking of platelets by fibrinogen and requires the activation of platelets plus the binding of fibrinogen. The extent of aggregation was assessed by PRU, determined by the VerifyNow P2Y12 assay. The VerifyNow P2Y12 assay is designed to directly measure the effects of drugs on the P2Y12 receptor, using prostaglandin E1 in addition to ADP to increase intraplatelet cAMP. Platelet reactivity was expressed in PRU.
Time Frame: as for outcome 2
Population: Participants treated with cangrelor and prasugrel or clopidogrel were used for the analysis and presentation of data.
Measure: Mean (Standard Deviation); unit: PRU
Groups:
- Prasugrel 30 Min After Cangrelor: Prasugrel 60 mg was administered orally 30 min after the discontinuation of cangrelor infusion (2.5 hrs after initiation of cangrelor infusion).
  Cangrelor IV was administered as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs on study Day 1.
- Clopidogrel Within 5 Min After Cangrelor: Clopidogrel 600 mg was administered orally within 5 min after the discontinuation of the cangrelor infusion (2 hrs after initiation of cangrelor infusion).
  Cangrelor IV was administered as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs on study Day 1.
- Clopidogrel 1.5 Hrs During Cangrelor: Clopidogrel 600 mg administered orally 1.5 hrs following the initiation of cangrelor infusion.
  Cangrelor IV was administered as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs on study Day 1.
- Clopidogrel 1 Hr During Cangrelor: Clopidogrel 600 mg administered orally 1 hr following the initiation of cangrelor infusion.
  Cangrelor IV was administered as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs on study Day 1.
Arm/Group | Prasugrel 30 Min After Cangrelor | Clopidogrel Within 5 Min After Cangrelor | Clopidogrel 1.5 Hrs During Cangrelor | Clopidogrel 1 Hr During Cangrelor
Number analyzed (Participants) | 3 | 3 | 6 | 3
PRU
  Cangrelor Reference (2.5, 2, 1.5, or 1 hrs) | 208.0 (30.2) | 7.3 (5.1) | 17.7 (18.2) | 7.0 (2.0)
  1.75 hrs | 3.3 (2.3) | 3.7 (2.1) | 25.0 (30.5) | 6.3 (1.5)
  2 hrs | 5.3 (2.1) | NA (NA) — Per protocol, analysis was not performed for this arm at 2 hrs. | 28.8 (18.2) | 5.7 (2.1)

5. Secondary Outcome: Bleeding Events In Accordance With GUSTO Scale
Description: Bleeding was assessed by history, physical exam, and complete blood count (CBC) that was performed on study Day 1. Reports of bleeding were to be evaluated by performance of a CBC. Participants were assessed for bleeding events in accordance with the Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) scale.
  The severity of bleeding events by GUSTO Criteria is defined as the following:
  * Severe/life-threatening: fatal, intracranial hemorrhage, or if hemodynamic compromise results
  * Moderate: transfusion required
  * Mild: no transfusion or hemodynamic compromise
  A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Screening through the follow-up period (5 to 7 days after Day 1)
Population: Safety Population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: bleeding events
Groups:
- Prasugrel 30 Min After Cangrelor: Prasugrel 60 mg was administered on Day 1 as a single oral dose 30 min after the discontinuation of cangrelor infusion (2.5 hrs after initiation of cangrelor infusion).
  Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
Arm/Group | Prasugrel 30 Min After Cangrelor | Clopidogrel Within 5 Min After Cangrelor | Clopidogrel 1.5 Hrs During Cangrelor | Clopidogrel 1 Hr During Cangrelor
Number analyzed (Participants) | 3 | 3 | 6 | 3
bleeding events
  Mild | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0
  Life-threatening/Severe | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening through the follow-up period (5 to 7 days after Day 1)
Groups:
- Clopidogrel 1 Hr During Cangrelor: Cangrelor IV was administered on Day 1 as a 30 μg/kg bolus, followed by 4 μg/kg/min infusion for 2 hrs.
  Clopidogrel 600 mg administered on Day 1 as a single oral dose 1 hr following the initiation of cangrelor infusion.
Arm/Group | Prasugrel 30 Min After Cangrelor | Clopidogrel Within 5 Min After Cangrelor | Clopidogrel 1.5 Hrs During Cangrelor | Clopidogrel 1 Hr During Cangrelor
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes